CLINICAL TRIAL: NCT06293443
Title: Evaluation of Functionality of Unilateral Lower Extremity Amputees Grouped According to the Medicare Functional K Classification System-Single Blind Study
Brief Title: Evaluation of Functionality of Amputees According to the Medicare Functional K Classification System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Tugba Tanis, Principal Investigator, Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMU-OP-TT-01
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Amputation; Amputation; Traumatic, Leg, Lower

STUDY DESIGN:
Masking Description: participants underwent functional testing at clinical centers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lower extremity unilateral amputee (Other): Unilateral transtibial and unilateral transfemoral amputees were evaluated in the study. Criteria for autees to participate in the study; Being a unilateral lower extremity amputee, using a prosthesis, being literate, being between the ages of 18-65, having a healthy stump, and using their current prosthesis in daily life activities. Individuals who had knee disarticulation amputation and individuals who had hip disarticulation amputation were not included in the study.
  Interventions: Other: Lower extremity unilateral amputee

INTERVENTIONS:
Other: Lower extremity unilateral amputee — To evaluate the functionality of lower extremity unilateral amputees, to ensure that the results of the Medicare Functional K Classification System, which provides subjective data for the evaluator, become an objective evaluation method and to determine the functional levels of unilateral amputees; To create an objective data set by applying one-leg standing test, Ten meter walking test, L test, figure-8 walking test, joint range of motion, amputee mobility estimator scale, Houghton scale and joint position sense evaluation tests.

SUMMARY:
The aim of our study is; To evaluate the functionality of lower extremity unilateral amputees, to ensure that the results of the Medicare Functional K Classification System, which provides subjective data for the evaluator, become an objective evaluation method and to determine the functional levels of unilateral amputees; To create an objective data set by applying one-leg standing test, ten meter walking test, L test, figure-8 walking test, joint range of motion, amputee mobility estimator scale, houghton scale and joint position sense evaluation tests.

DETAILED DESCRIPTION:
The study will be carried out at Medicom Orthosis Prosthesis Center and Ortoport Prosthesis Application Center. The study will be conducted in accordance with the principles of human experimentation as defined in the Declaration of Helsinki. For this purpose, amputees who will participate in the study will be given detailed information about the study and will have to sign an informed consent form. 20 unilateral lower extremity amputations will be taken. The inclusion and exclusion criteria of the study are as follows; Inclusion criteria;

Unilateral lower extremity amputation, Using a prosthesis, Being literate, Being between the ages of 18-65, Having a healthy stump, Using your current prosthesis in daily living activities,

Exclusion criteria; Bilateral lower extremity amputation, Unilateral or bilateral amputation of the upper extremity, Having a cognitive or mental problem, Having serious hearing and vision problems, The individual has an orthopedic disease other than amputation, Having an uncontrolled neurological and systemic systemic disease,

SPPS 25.0 (Statistical Package for the Social Sciences) statistical package program will be used to evaluate the data. When the differences between two groups are desired to be evaluated, "Student's t Test" is used if it meets the parametric test prerequisites; If not, the "Mann Whitney-U test" will be used.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lower extremity amputation,
* Being using a prosthesis,
* Being literate,
* Being between the ages of 18-65,
* Having a healthy stump,
* Using your current prosthesis in daily living activities,

Exclusion Criteria:

* Bilateral lower extremity amputation
* Unilateral or bilateral amputation of the upper extremity,
* Having a cognitive or mental problem,
* Having serious hearing and vision problems,
* The individual has an orthopedic disease other than amputation,
* Having an uncontrolled neurological and systemic systemic disease,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Amputee Mobility Scale | 2 weeks
  It is a 21-item scale that evaluates static and dynamic balance. It is also used to predict the amputee's potential ambulation level. It is also a scale used to evaluate function during or after rehabilitation. Questions include sitting balance, transfers, standing balance, walking, stairs, assistive device use. Scoring is made between 0-47.

SECONDARY OUTCOMES:
One Leg Standing Test | 2 weeks
  This test measures balance and standing ability. It is done by keeping time. The patient is asked to stand on one leg with arms at either side of the body. The test is performed in two ways, with eyes open and closed. The patient is asked to lift one leg up while standing. If the patient is using an assistive device such as a cane, the time is recorded when the patient stops holding it, or when the patient lifts his foot up. The time is stopped when the patient's foot touches the ground. If a loss of balance occurs in less than 5 seconds, the test is terminated. If the patient can stand on one leg for 30 seconds, the test is said to be over. If the cut-off value is <10 seconds, there is a balance disorder; if it is <5 seconds, there is a risk of falling. The score in the test is related to age and as age increases, the score decreases.
Houghton Scale | 2 weeks
  It is a scale that objectively evaluates the level of independence of lower extremity amputees with their prostheses. The scale parallels the Medicare Functional K Classification System. A Houghton Scale score ≥ 9 corresponds to a level K3 or K4 amputee, Houghton Scale scores 6-8 correspond to a level K2 amputee, and a Houghton Scale score ≤ 5 corresponds to a level K1 amputee. The Houghton scale is a scale scored between 0-12.
8-Shape Walking Test | 2 weeks
  It is one of the tests that measures speed and agility abilities together. It measures the daily walking ability of older adults with mobility impairments (8). 8ŞYT tests a participant's walking on both straight and curved paths. It uses a path in which the participant is asked to walk in a figure eight around two cones. Scores are recorded in two areas: speed (time to complete), amplitude (number of steps taken).
joint range of motion | 2 weeks
  The presence of limitation will be evaluated by checking the normal joint movements of the amputees, and whether there is an effect on the ROM values during the use of the prosthesis will be taken into account. Joint range of motion of amputees will be evaluated using the Goniometer-Pro smartphone application.
  Joint range of motion will be measured based on reference and pivot points in supine and prone positions. Measurements will be taken on both sides and noted. In unilateral transtibial amputee; Range of motion in knee joint flexion, extension, hip joint flexion, extension and trunk flexion, extension and lateral flexion will be checked. In unilateral transfemoral amputee; Hip joint flexion, extension and trunk flexion, extension, lateral flexion range of motion will be measured based on standing reference and pivot points. Measurements will be taken on both sides and noted.
proprioception | 2 weeks
  With this test, joint position sense, which is a component of proprioception, will be measured. Joint position sense is a person's ability to perceive the position sense of a joint and restore it when the position of the extremity is changed. The most well-known tests in the evaluation of proprioception measure the person's capacity to actively or passively perform a targeted joint position (active/passive repositioning test) or the threshold of perceiving the desired joint movement (movement detection threshold test).
l test | 2 weeks
  It is a performance-based measure that can be used to evaluate physical function, including dynamic balance ability. The test is a modification of the "Timed Up and Go" test. The L-test allows evaluation of walking over a longer walking distance and involves turning in two directions. Amputees have a 1-minute rest period between trials and a 2-minute rest period between measurements. Amputees are instructed to walk at comfortable walking speeds, with or without their usual walking aids. Before participation, a standard demonstration and explanation of both outcome measures is given. In order to perform the test; 1 stopwatch, 1 chair, 3 meters and 7 meters long walking area are required.
10 Meter Walking Test | 2 weeks
  It is a test that evaluates the walking performance of an amputee. This test is a performance test used to evaluate walking speed over a short distance in meters per second. The equipment required for the test is a stopwatch and a ground with a specified distance. Total time for scoring is recorded in meters/second. An individual assistive device may be used, but must be kept consistent and documented for each test. Three trials are made and the average of these three trials is taken. Patients are asked to walk a distance of 10 meters in a straight line on a flat road, at their own pace, using assistive walking devices, if any.

CONTACTS AND LOCATIONS:
Overall Officials: GİZEM BOZTAŞ ELVERİŞLİ, Study Director — Medipol University
Locations (1):
- Istanbul Medıpol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No